CLINICAL TRIAL: NCT04581109
Title: Detection of Viable CTCs Using the EPIDROP Technology in Metastatic Prostate Cancer
Brief Title: Detection of Viable CTCs Using the EPIDROP Technology in Metastatic Prostate Cancer (EPIDROP)
Acronym: EPIDROP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL17_0318; 2018-A03249-46 (Other: ANSM)
Record Dates: First submitted 2020-10-02; First posted 2020-10-09 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Circulating tumor cells (CTCs); Biomarker; CellSearch; EPIDROP
MeSH Terms: conditions — Prostatic Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with metastatic prostate cancer (Experimental)
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Twenty ml of blood will be drawn from each patient : 10 ml of blood will be drawn on CellSave tubes (fixed cells) for CTC detection using the FDA-cleared CellSearch system (gold standard) and 10 ml of blood will be drawn on EDTA tubes (viable cells) for the detection of functional CTCs using the EPIDROP.

SUMMARY:
The use of liquid biopsy could be the key for precision medicine. Circulating tumor cells (CTCs) are the most studied circulating biomarkers used to assess the metastatic process and they have shown their clinical validity and utility in cancer patients. However, their detection and capture are still a challenge as they are very rare in the bloodstream. In this clinical trial named "EPIDROP", the investigators will use an innovative device called EPIDROP (for EPIspot in a DROP) in metastatic prostate cancer. EPIDROP is a completely new technology answering to biological and clinical questions by proposing a procedure detecting the functional subset of prostatic CTCs at the single cell level. The investigators will stain cells in the sample for EpCAM, PSMA, CD45 before to encapsulate them one by one in microdroplets and measure the PSA secretion by only the viable CTCs. This study aims to demonstrate the non-inferiority of the EPIDROP compared to the CellSearch system.

DETAILED DESCRIPTION:
Methods :

One hundred patients with a metastatic prostate cancer will be recruited plus 50 healthy donors. Twenty ml of blood will be drawn : 10 ml of blood will be drawn on CellSave tubes (fixed cells) for CTC detection using the FDA-cleared CellSearch system (gold standard) and 10 ml of blood will be drawn on EDTA tubes (viable cells) for the detection of functional CTCs using the EPIDROP. Patients will be followed for 18 months.

Samples from fifty control subjects will be provided by the Etablissement Français du Sang.

ELIGIBILITY:
Inclusion Criteria :

* To be male, over 18 years old
* Metastatic prostate cancer naive to any treatment or metastatic prostate cancer in biological recurrence (PSA increase) and/or clinical recurrence after hormone suppression (mCRPC)

Exclusion Criteria:

* Non-metastatic prostate cancer in biological and/or clinical recurrence after hormone-suppression (nmCRPC)
* Other active or treated cancer less than 5 years old
* Be protected by law (guardianship or curatorship)
* Be deprived of liberty by administrative decision
* Not being affiliated to a social security scheme, or not being a beneficiary of such a plan
* Being in a period of exclusion from another protocol
* Inability to understand and/or respond to questionnaires
* Inability to understand the nature, purpose and methodology of the study
* Refusal to sign informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
EPIDROP technique sensitivity versus CellSearch system sensitivity | At 18 months
  Proportion of true positive and false negative patients with a confidence interval
EPIDROP technique specificity versus CellSearch system specificity | At 18 months
  Proportion of true negative and false positive healthy controls with a confidence interval

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital Center, Montpellier, Occitanie
  - University Center, Hospital, Nîmes

IPD SHARING:
Plan to Share IPD: No